CLINICAL TRIAL: NCT07268508
Title: Randomised Controlled Trial Evaluating the Impact of a Pro-diversity Gut Microbiota Diet on Gut Microbiota, Eating Behaviour and Sensory Function in Patients Who Have Undergone Bariatric Surgery
Brief Title: Impact of a Pro-diversity Gut Microbiota Diet After a Bariatric Surgery on Gut Microbiota, Eating Behaviour and Sensory Function
Acronym: BariaGut Taste
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 69HCL24_0033
Record Dates: First submitted 2025-08-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Obesity (Disorder); Bariatric Surgery
Keywords: Bariatric surgery; gut microbiota; sensory alteration; food preferences; weight loss maintenance
MeSH Terms: conditions — Obesity; Food Preferences | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: * Arm with nutritional counselling promoting gut microbiota diversity
  * Arm with standard nutritional counselling
Who Masked: Participant
Masking Description: Randomisation will be stratified according to sex, type of surgery and age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with nutritional counselling promoting gut microbiota diversity (Experimental): Given the low amounts of food consumed during the first months after surgery, the specific nutritional recommendations for this group will be implemented starting 3 months post-surgery. Before 3 months, participants will receive the standard nutritional recommendations of routine care after bariatric surgery, identical to those given to the second group (see below).
  From 3 months onwards, participants will be encouraged to increase the consumption of certain specific foods known for their benefits on the gut microbiota, particularly for promoting gut bacterial diversity, in addition to maintaining protein intake and paying attention to food textures. Summary sheets will be provided to help recall the recommendations.
  Interventions: Other: Nutritional counseling
- Participants with standard nutritional counselling (No Intervention): The nutritional recommendations given to participants in this group are those applied in routine care within the Endocrinology, Diabetes, and Nutrition (EDN) Department for patients who have undergone sleeve gastrectomy or gastric bypass (Roux-en-Y).
  These recommendations aim to maintain adequate protein intake and are adapted to the recent changes in their digestive tract (pureed then mashed food during the first postoperative month). During the first 6 months, patients' food intake is significantly below their nutritional needs. So it is important to pay close attention to hydration (away from meals) and macronutrient intake, especially proteins, as well as the progression of food texture and chewing.

INTERVENTIONS:
Other: Nutritional counseling — Nutritional counseling
  Arms: Participants with nutritional counselling promoting gut microbiota diversity

SUMMARY:
Bariatric surgery is the most effective treatment for long-term weight loss and reducing obesity-related health risks. It alters the gastrointestinal tract as well as metabolic and hormonal functions, influencing eating behaviour. However, weight loss outcomes and long-term maintenance vary between patients, likely due to changes in the gut microbiota. Dietary recommendations aimed at improving microbiota diversity could help support sustained weight loss after surgery.

The BariaGut Taste study aims to compare two dietary approaches following bariatric surgery: nutritional counselling promoting gut microbiota diversity versus standard nutritional counselling. One year after surgery, the study will evaluate differences in microbiota diversity, changes in food preferences and eating behaviours, sensory profiles (taste, smell), levels of digestive and gut hormones fasting, before and after eating, cardiometabolic parameters, mental health, physical activity, and more, to better understand Bariatric surgery is the most effective treatment for long-term weight loss and reducing obesity-related health risks. It alters the gastrointestinal tract as well as metabolic and hormonal functions, influencing eating behaviour. However, weight loss outcomes and long-term maintenance vary between patients, likely due to changes in the gut microbiota. Dietary recommendations aimed at improving microbiota diversity could help support sustained weight loss after surgery.

The BariaGut Taste study aims to compare two dietary approaches following bariatric surgery: nutritional counselling promoting gut microbiota diversity versus standard nutritional counselling. One year after surgery, the study will evaluate differences in microbiota diversity, changes in food preferences and eating behaviours, sensory profiles (taste, smell), levels of digestive and gut hormones fasting, before and after eating, cardiometabolic parameters, mental health, physical activity, and more, to better understand the mechanisms that may explain variations in response to bariatric surgery.

The BariaGut Taste study is a prospective, randomized, controlled trial with two parallel groups, involving non-diabetic patients aged 25 to 65 y undergoing either sleeve gastrectomy or Roux-en-Y gastric bypass. The trial will be conducted at the digestive surgery department of Edouard Herriot Hospital, the endocrinology-diabetes-nutrition department of Lyon Sud Hospital Center, and the Human Nutrition Research Center Rhône-Alpes. 60 participants are expected to be recruited, with 30 in each arm.

Participants will be enrolled before surgery during a routine care visit with the surgeon. They will then undergo a metabolic assessment visit conducted exclusively for research purposes. This visit will allow to collect baseline data on primary outcomes via blood, expired air, and stool samples, anthropometric measurements, indirect calorimetry, a battery of questionnaires (TFEQ-21, DEBQ, PHQ-9, SF36, GSES, PANAS, ESUL, BES, DERS, GAD-7, IPAQ, BAQ, GSRS, sensory alterations, Bristol and Likert scales, and FNS), computerized food preference tests (LFPQ), and a standardized, video-recorded ad libitum buffet.

Participants will be followed up at 3, 6, and 12 months after surgery through visits combining clinical care and research assessments. The dietary interventions specific to each group will be provided since the 3-month visit. The assessments conducted before surgery will be repeated at 6 and 12 months, also integrating clinical care objectives.

Additional blood, stool, and adipose tissue samples collected during surgery will be stored to create a biobank.

ELIGIBILITY:
Inclusion Criteria:

* Between 25 and 65 years old
* Undergoing either sleeve gastrectomy or Roux-en-Y gastric bypass
* With grade 3 obesity (BMI≥40 kg/m²) or with BMI≥35 kg/m² and at least one comorbidity likely to be improved after surgery, with the exception of type 2 diabetes
* Signed consent form
* Living less than an hour and 30 minutes from the hospital
* Presence of effective and stable contraception for women of childbearing potential

Exclusion Criteria:

* Type 2 diabetes
* Presence of a contraindication to bariatric surgery
* Presence of gastrointestinal pathologies with an inflammatory component, known gastroparesis, total gastrectomy, colectomy, exocrine pancreatic insufficiency, known endocrine pathologies inducing hyperglycaemia (uncontrolled dysthyroidism, acromegaly, hypercorticism, etc.), severe chronic renal insufficiency (< 30mL/min), or hepatocellular insufficiency
* Claustrophobic
* Pregnant or breastfeeding women
* Taking an obesity treatment 3 months before surgery
* Taking a corticoids, immunosuppression, anabolizing, or growing hormones, antibody treatments less than 3 months before inclusion
* Daily taking of laxatives or drugs that can strongly interfere with the composition of the intestinal microbiota. If taken sporadically, the patient can be included at a distance (3 weeks) from the laxatives taken.
* Specific diets (vegetarian, vegan or without gluten)
* No French speaker
* Already included in other study
* Donated blood in the last two months
* Without freezer access
* With allergy or intolerance to food propose in ad libitum buffet

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Microbiota diversity 12 months after surgery | Primary outcome will be assessed three times : before the surgery, 6 and 12 months after
  The change in the diversity of the microbiota (shot gun metagenomic analysis, counting the number of microbial genes), between before surgery and one year after surgery (delta) between the two dietary intervention groups.

SECONDARY OUTCOMES:
Eating behaviour during a standardised, filmed and validated ad libitum buffet : Food intake | Before the surgery and at 6 and 12 month after
  energy intake, macro- and micronutrient intake The items chosen during the buffet from the 17 items that will be offered will be noted. The quantities in g and calories consumed of each item will be estimated from the weighing of the plates before and after the buffet, the contribution of each of the items to the energy intake will also be evaluated.
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Nutritional quality | Before the surgery and at 6 and 12 month after
  Nutritional quality through analysis of the foods chosen and consumed Buffet items are classified (pre-defined classification) into seven groups based on their macronutrient content and energy density: starchy foods, meat and fish, fruits and vegetables, dairy products, sweet desserts, sauces, and sweetened beverages. They are also classified according to their fat, sugar, and protein content, and their energy density (4 groups).
  The quantities consumed in grams and as a percentage of energy intake per group will be assessed for each subject and per visit.
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  time spent selecting food at the buffet, duration of ingestion, ingestion speed, total meal duration, number of bites per minute, total number of bites and bites by food type, and food choices
  Several indicators will be assessed for the buffet's microstructure based on the analysis of videos taken during the buffet:
  - Buffet time
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal appreciation | Before the surgery and at 6 and 12 month after
  time spent selecting food at the buffet, duration of ingestion, ingestion speed, total meal duration, number of bites per minute, total number of bites and bites by food type, and food choices Assessed with visual analog scale from 1(worse outcome) to 10 (better outcome)
Eating behaviour and preferences : Behaviors | Before the surgery and at 6 and 12 month after
  binge eating using sub-scores from tthe BES (Binge Eating Scale) for binge eating
  BES : Binge Eating Scale - score from 0 to 46, score of 46 = highest level of binge eating disorder
Eating behaviour and preferences : Food preferences | Before the surgery and at 6 and 12 month after
  Food preferences using the short version of the LFPQ (Leeds Food Preference Questionnaire) LFPQ : Leeds Food and Preference Questionnaire- score from 0 to 100 on preference or motivation for a type of food, high score = strong preference or motivation
Appetite : hunger level | Before the surgery and at 6 and 12 month after
  Assessed using visual analog scales rated from 0 (worse outcome) to 10 (better outcome) on the following dimensions : hunger
Appetite : satiety | Before the surgery and at 6 and 12 month after
  Assessed using visual analog scales rated rom 0 (worse outcome) to 10 (better outcome) on the following dimensions : feeling of satiety
Appetite : desire to eat | Before the surgery and at 6 and 12 month after
  Assessed using visual analog scales rated from 0 (worse outcome) to 10 (better outcome) on the following dimensions : desire to eat
Appetite : prospective consumption | Before the surgery and at 6 and 12 month after
  Assessed using visual analog scales rated from 0 (worse outcome) to 10 (better outcome) on the following dimensions : consommation
Appetite : meal appreciation | Before the surgery and at 6 and 12 month after
  Assessed using visual analog scales rated rom 0 (worse outcome) to 10 (better outcome) on the following dimensions : meal appreciation
Sensory functions : detection scores | Before the surgery and at 6 and 12 month after
  Assessed using Taste Strips tests
Sensory functions : intensity | Before the surgery and at 6 and 12 month after
  Assessed using Taste Strips tests
Sensory functions : pleasantness | Before the surgery and at 6 and 12 month after
  Assessed using Taste Strips tests
Sensory functions : edibility of tastes | Before the surgery and at 6 and 12 month after
  Assessed using Taste Strips tests
Sensory functions : edibility of odors | Before the surgery and at 6 and 12 month after
  Assessed using Taste Strips tests
Self-reported alterations in sensory functions | Before the surgery and at 6 and 12 month after
  Assessed using dedicated questions
Body perception | Before the surgery and at 6 and 12 month after
  Assessed using the BAQ questionnaire (Body Awareness Questionnaire) BAQ : Body Awarness Questionnaire - score from 13 to 65, score of 65 = positive assessment of one's body
Appetite : desire to eat | Before the surgery and at 6 and 12 month after
  Assessed using visual analog scales rated from 0 to 10 on the following dimensions: desire to eat
Appetite : prospective consumption | Before the surgery and at 6 and 12 month after
  Assessed using visual analog scales rated from 0 to 10 on the following dimensions
Microbiota composition | Before the surgery and at 6 and 12 month after
  Evaluated via gene function analysis from metagenomics data, metabolomics and short-chain fatty acid quantification
Microbiota function | Before the surgery and at 6 and 12 month after
  Evaluated via gene function analysis from metagenomics data, metabolomics and short-chain fatty acid quantification
Endocrine, digestive or intestinal hormones | Before the surgery and at 6 and 12 month after Fasting (all except acylated ghrelin), before the buffet and 1 hour after (adiponectin, total GLP1, ghrelin, acylated ghrelin, total PYY, glucagon, GIP and FGF-19)
  Blood sample to measure :
  Adiponectin µg/ml
Exhaled gas profiles | Before the surgery and at 6 and 12 month after
  Assessed by volatolomic signatures
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  BMI will be assessed
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  Energy metabolism by indirect calorimetry
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  postprandial plasma markers: We will assess: glycaemia (g/L)
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  CRP
Vital parameters | Before the surgery and at 6 and 12 month after
  Blood pressure
Nutritional status: Blood vitamin | Before the surgery and at 6 (except plasma fatty acid profile) and 12 month after
  Blood vitamin status :
  For the research, we will focus only whether or not the participant has a deficiency in one of the vitamins measured (yes/no variable).
  The vitamins assessed are :
  - Vitamin B12 (pmol/L) should be above 145 pmol/L
Nutritional status : Blood mineral | Before the surgery and at 6 (except plasma fatty acid profile) and 12 month after
  Blood mineral status:
  * Calcium (mmol/L) should be above 64 mmol/L
  * Phosphor (mmol/L) should be above 0.81 mmol/L
  * Magnesium (mmol/L) should be above 0.66 mmol/L
  * Sodium (mmol/L) should be above 136 mmol/L
  * Potassium (mmol/L) should be above 3.4 mmol/L
  * Chlore (mmol/L) should be above 98 mmol/L
Nutritional status : Plasma fatty acid | Before the surgery and at 6 (except plasma fatty acid profile) and 12 month after
  Plasma fatty acid profile
Nutritional status : Protein | Before the surgery and at 6 (except plasma fatty acid profile) and 12 month after
  Protein status
Average energy | Before the surgery and at 6 and 12 month after
  Assessed using 3-day dietary recall randomly selected from the 7 days preceding the visits
macronutrients intakes and proportions | Before the surgery and at 6 and 12 month after
  Assessed using 3-day dietary recall randomly selected from the 7 days preceding the visits
micronutrients intakes and proportions | Before the surgery and at 6 and 12 month after
  Assessed using 3-day dietary recall randomly selected from the 7 days preceding the visits
Mental health: Quality of life | Before the surgery and at 6 and 12 month after
  Quality of life using the SF36 questionnaire SF36 - health status questionnaire - score from 0 to 100, score of 100 = excellent perceived health
Mental health: Self-confidence | Before the surgery and at 6 and 12 month after
  Self-confidence and self-efficacy using the GSES GSES: Generalized Self-Efficacy Scale - score of 10 to 40, score of 40 = strong confidence in one's ability to effectively manage different life situations and challenges
Mental health: Depression | Before the surgery and at 6 and 12 month after
  Depression with PHQ-9 PHQ-9: Patient Health Questionnaire
  -score from 0 to 27, score of 27=severe depression
Mental health: Anxiety | Before the surgery and at 6 and 12 month after
  Anxiety assessment using GAD-7 GAD-7: Generalized Anxiety Disorder - if score >7 then anxiety disorders should be suspected
Physical activity | Before the surgery and at 6 and 12 month after
  Assessed using the short version of the IPAQ IPAQ: International Physical Activity Questionnaire - continuous daily energy expenditure score, high score means high AP
  The questionnaire allows the subject to be classified according to 3 levels of activity: inactive, moderate, high.
Emotions: positive and negative | Before the surgery and at 6 and 12 month after
  positive and negative emotion assessed using the PANAS scale PANAS: Positive Affectivity and Negative Affectivity Scale - 2 scores from 10 to 50 - positive affectivity score = 50 best, negative affectivity score = 50 worst
Emotions: food phobias | Before the surgery and at 6 and 12 month after
  food phobias using the FNS questionnaire FNS : Food Neophobia Scale -score from 10 to 70 - score of 70 = neophobia, i.e. less willingness to try new foods
Emotions: loneliness | Before the surgery and at 6 and 12 month after
  loneliness using the ESUL questionnaire University of Laval Loneliness Scale - score from 20 to 80, score of 80 = most pronounced feeling of loneliness
Changes in stool consistency | Before the surgery and at 6 and 12 month after
  Assessed using Bristol stool scale Bristol scale : 7 types of stools to choose from photo: type 1 = hard and lumpy stools, type 7 = completely liquid stools
Changes in stool frequency | Before the surgery and at 6 and 12 month after
  Assessed using Bristol stool scale : 7 types of stools to choose from photo: type 1 = hard and lumpy stools, type 7 = completely liquid stools
Changes in gastrointestinal symptoms | Before the surgery and at 6 and 12 month after
  Assessed using Bristol stool scale
Grade of hepatic steatosis | Before the surgery and at 12 month after
  Evaluation by FibroScan® but only for patients who had a FibroScan® performed before surgery.
Grade of hepatic fibrosis | Before the surgery and at 12 month after
  Evaluation by FibroScan® but only for patients who had a FibroScan® performed before surgery.
Eating behaviour and preferences : Behaviors | Before the surgery and at 6 and 12 month after
  Behaviors (emotional eating and cognitive restraint) using score from the DEBQ (Dutch Eating Behavior Questionnaire) a DEBQ : Dutch Eating Behaviour Questionnaire : 3 sub-scores: cognitive restriction, reactivity to external stimuli and emotionality from 1 to 5, score 5 = strong impact of eating behavior
Hepatic metabolic flexibility | Before the surgery and at 6 and 12 month after
  Assessed via the degree of alteration of MAMs (Mitochondia-Associated Membranes) in peripheral blood mononuclear cells (PBMCs), only for patients who had a FibroScan® performed before surgery.
Safety parameters | Before the surgery and at 6 and 12 month after
  thyroid function: Thyroid function is assessed based on TSH levels in mIU/L (should be above 0.4 mIU/L and below 4.8 mIU/L), 2.
  The assessment for the research is whether the measures are within the limits or not (yes/no variable).
Compliance and follow-up of advice given during the intervention | until month 12
  Based on the three 24-hour reminders completed by participants before each visit, the dietitian will classify participants into three categories: good, average or poor compliance.
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  time spent selecting food at the buffet
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  duration of ingestion
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  ingestion speed
Changes in stool consistency | Before the surgery and at 6 and 12 month after
  Assessed using Likert scale Likert scale : 7 types of stools to choose from photo: type 1 = hard and lumpy stools, type 7 = completely liquid stools
Changes in stool consistency | Before the surgery and at 6 and 12 month after
  Assessed using gastrointestinal symptoms using GSRS Gastrointestinal Symptom Questionnaire - score 15 to 105, score 105=severe gastrointestinal symptoms
Safety parameters | Before the surgery and at 6 and 12 month after
  complete blood count
Safety parameters | Before the surgery and at 6 and 12 month after
  AST
Safety parameters | Before the surgery and at 6 and 12 month after
  ALT
Safety parameters | Before the surgery and at 6 and 12 month after
  gamma GT
Safety parameters | Before the surgery and at 6 and 12 month after
  bilirubin
Safety parameters | Before the surgery and at 6 and 12 month after
  alkaline phosphate
Safety parameters | Before the surgery and at 6 and 12 month after
  creatinine
Safety parameters | Before the surgery and at 6 and 12 month after
  uric acid
Safety parameters | Before the surgery and at 6 and 12 month after
  ionogram results: Sodium (mmol/L) which should be between 136 and 145 Potassium (mmol/L) which should be between 3.4 and 4.5 Chlorine (mmol/L) which should be between 98 and 107 Bicarbonates (mmol/L) which should be between 22 and 29
Safety parameters | Before the surgery and at 6 and 12 month after
  coagulation : prothrombin time
Changes in stool frequency | Before the surgery and at 6 and 12 month after
  Assessed using Likert scale
Changes in stool frequency | Before the surgery and at 6 and 12 month after
  Assessed using gastrointestinal symptoms using GSRS : 15 questions with answers from No discomfort at all at Very severe discomfort (7 levels)
Changes in gastrointestinal symptoms | Before the surgery and at 6 and 12 month after
  Assessed using Likert scale
Changes in gastrointestinal symptoms | Before the surgery and at 6 and 12 month after
  gastrointestinal symptoms using GSRS
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  total meal duration
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  number of bites per minute
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  total number of bites
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  bites by food type
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  food choices
Eating behaviour during a standardised, filmed and validated ad libitum buffet: Meal microstructure | Before the surgery and at 6 and 12 month after
  Calorie intake consumed per minute of the buffet
Safety parameters | Before the surgery and at 6 and 12 month after
  ionogram results:
  Anion gap = (Na+ + K+) - (HCO3- + Cl-) (mmol/L) which should be between 12 and 20
Endocrine, digestive or intestinal hormones | Before the surgery and at 6 and 12 month after Fasting (all except acylated ghrelin), before the buffet and 1 hour after (adiponectin, total GLP1, ghrelin, acylated ghrelin, total PYY, glucagon, GIP and FGF-19)
  Blood sample to measure :
  Ghrelin pg/ml acylated ghrelin pg/ml
Endocrine, digestive or intestinal hormones | Before the surgery and at 6 and 12 month after Fasting (all except acylated ghrelin), before the buffet and 1 hour after (adiponectin, total GLP1, ghrelin, acylated ghrelin, total PYY, glucagon, GIP and FGF-19)
  Blood sample to measure :
  GIP pmol/l total GLP-1 : pmol/L glucagon : pmol/L
Endocrine, digestive or intestinal hormones | Before the surgery and at 6 and 12 month after Fasting (all except acylated ghrelin), before the buffet and 1 hour after (adiponectin, total GLP1, ghrelin, acylated ghrelin, total PYY, glucagon, GIP and FGF-19)
  Blood sample to measure :
  total PYY : ng/L
Endocrine, digestive or intestinal hormones | Before the surgery and at 6 and 12 month after Fasting (all except acylated ghrelin), before the buffet and 1 hour after (adiponectin, total GLP1, ghrelin, acylated ghrelin, total PYY, glucagon, GIP and FGF-19)
  Blood sample to measure :
  leptin : ng/ml
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  We will assess: insulin (mU/L)
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  We will assess: triglycerides (mmol/L), HDL (mmol/L), LDL (mmol/L), ApoB (mmol/L), sphingolipid (mmol/L) and unesterified fatty acid(mmol/L)
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  we will calculate: HOMA-IR (=insulin*glycarmia/22.5) and the total cholesterol/HDL cholesterol ratio.
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  postprandial plasma markers: We will assess: insulin (mU/L)
Nutritional status: Blood vitamin | Before the surgery and at 6 (except plasma fatty acid profile) and 12 month after
  Blood vitamin status :
  For the research, we will focus only whether or not the participant has a deficiency in one of the vitamins measured (yes/no variable).
  The vitamins assessed are :
  - Vitamin B9 (mmol/L) should be above 10.4 mmol/L
Nutritional status: Blood vitamin | Before the surgery and at 6 (except plasma fatty acid profile) and 12 month after
  Blood vitamin status :
  For the research, we will focus only whether or not the participant has a deficiency in one of the vitamins measured (yes/no variable).
  The vitamins assessed are :
  - Vitamin B1 (nmol/L) should be above 78 nmol/L
Nutritional status: Blood vitamin | Before the surgery and at 6 (except plasma fatty acid profile) and 12 month after
  Blood vitamin status :
  For the research, we will focus only whether or not the participant has a deficiency in one of the vitamins measured (yes/no variable).
  The vitamins assessed are :
  * Vitamin C (µmol/L) should be above 25 µmol/L
  * Vitamin A (µmol/L) should be above 1.40 µmol/L
Nutritional status : Blood mineral | Before the surgery and at 6 (except plasma fatty acid profile) and 12 month after
  Blood mineral status:
  * Iron (µmol/L) should be above 5.8µmol/L
  * Selenium (µmol/L) should be above 56µmol/L
  * Zinc (µmol/L) should be above 9.20µmol/L
Safety parameters | Before the surgery and at 6 and 12 month after
  thyroid function: Thyroid function is assessed based on free thyroxine in pmol/L (should be above 11.9 pmol/L and below 21.9 pmol/L)
  The assessment for the research is whether the measures are within the limits or not (yes/no variable).
Safety parameters | Before the surgery and at 6 and 12 month after
  thyroid function: Thyroid function is assessed based on free triiodothyronine in pmol/L (should be above 3.1 pmol/L and below 6.8 pmol/L).
  The assessment for the research is whether the three measures are within the limits or not (yes/no variable).
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  Waist-to-hip ratio will be assessed
Vital parameters | Before the surgery and at 6 and 12 month after
  resting heart rate
Safety parameters | Before the surgery and at 6 and 12 month after
  coagulation : activated partial thromboplastin time
Safety parameters | Before the surgery and at 6 and 12 month after
  coagulation : fibrinogen
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  We will assess: total cholesterol (g/L)
Cardio-metabolic profile parameters | Before the surgery and at 6 and 12 month after
  We will assess: HbA1c (mmol/mol),

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hospital Edouard Herriot, digestive surgery department, Lyon
  - Centre de recherche en nutrition humaine de Rhône-Alpes, Pierre-Bénite
  - Hôpital Lyon sud, Endocrinology Diabetes Nutrition department, Pierre-Bénite